CLINICAL TRIAL: NCT07268378
Title: Efficacy of Supervision of Oncology/Haematology Clinicians by Psycho-oncologists: A Randomized Controlled Trial
Brief Title: Supervision of Clinicians in Oncology by Psycho-oncologists : Evaluation
Acronym: SCOPE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Principal Investigator, Friedrich Stiefel, Head of Psychiatric Liaison Service, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SCOPE; KLS-6188-08-2024 (Other Grant/Funding Number: Ligue suisse contre le cancer)
Record Dates: First submitted 2025-09-02; First posted 2025-12-05 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Healthy Participants
Keywords: supervision; clinician; oncology; hematology; formative function; restorative function; normative function; reflexivity; feelings towards patients; burnout
MeSH Terms: conditions — Neoplasms; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in an intervention (Supervision group: SPV) group with supervision sessions and a waiting-control (CTRL) group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervision group (SPV) (Experimental): As baseline assessments (T0), participants will complete the Maslach Burnout Inventory (MBI) and 5-day clinical situation recordings (measuring supervisee's reflexivity) in which they describe a clinical situation that has remained in their mind during the day.
  Each participant will then take part in four 60 min clinician-centred supervision sessions (bi-monthly supervisions). During each supervision, (i) clinicians' feelings toward the patients presented will be measured with the Feeling Word Checklist (FWC-58) at the beginning and end of each session, and (ii) specific aspect and the overall quality of the supervision wil be assessed with a 4-item ad-hoc questionnaire for both supervisee and the supervisor.
  Assessments performed at T0 will be repeated after the 2-month intervention (T1). Finally, the MBI will be administered at follow-up assessments 3 months (FU3) and 6 months (FU6) after T1.
  Interventions: Other: Supervision session
- Waiting-control group (CTRL) (No Intervention): As baseline assessments (T0), participants will complete the Maslach Burnout Inventory (MBI) and 5-day clinical situation recordings (measuring supervisee's reflexivity). The clinical situation recordings consist of describing a clinical situation that has remained in the clinician's mind during the day.
  They will then not receive supervisions during the 2-month waiting period.
  Assessments will be repeated after the 2-month waiting period (T1: MBI and 5-day clinical situation recordings) and follow-up evaluations with the MBI will take place at 3 months (FU3) and 6 months (FU6).
  After the trial period (i.e., after FU6), participants in this arm will be offered the opportunity to reveice the intervention.

INTERVENTIONS:
Other: Supervision session — In the first and thrid sessions, supervisees will comprehensively describe a clinical situation with a patient, which strongly affected them in a very negative way (e.g., feelings of rejection, anxiety, anger), or even lead to words (e.g., outbursts, impoliteness, cynicism) and actions (e.g., avoidance of the patient, forgetting appointments, deviation from good medical practice).
  In the second and fourth sessions, the same proceeding takes place, with the exception that participants are invited to present a clinical encounter with a patient, which strongly affected them in a very positive way (e.g., feelings of intense closeness, sympathy, pronounced mourning after the patient's death), or even lead to words (e.g., self-disclosure, discussing private information, compliments) and actions (e.g., special favours, difficulties to end treatment, deviation from good medical practice).
  Arms: Supervision group (SPV)

SUMMARY:
Communication in the oncology setting involves cognitive as well as emotional challenges for both clinicians and patients, and interactional dimensions that emerge in their encounter. Supervision of oncology/haematology clinicians by psycho-oncologists is one of the most frequently used tools, which aims to enhance their communicative and relational competences, and at the same time to support them in their daily clinical work. However, little is known regarding its impact and how the supervisory process acts upon clinicians. This study thus aims to evaluate the efficacy of four 1-hour supervision sessions following a clinician-centred format, which allows supervisors to rapidly access supervisees' own difficulties in the encounter with certain patients. In addition, the supervisory process will be examined qualitatively by analysing in-depth audio-taped supervision sessions. The focus of analysis will be "what works" and "what does not". If beneficial effects are found, clinician-centred supervision -- thanks to its focused and time saving format -- could be realistically implemented for nurses and physicians working in the oncology and haematology settings. Effects are expected on clinicians' capacity to reflect on challenging encounters with patients, on potential negative feelings towards patients, and on clinicians' professional well-being. The clinician-centred supervision format could be easily taught to psycho-oncologists who wish to start supervising haematology and oncology clinicians. Clinicians who are less preoccupied with themselves, or with negative feelings towards their patients, have more supportive relationships with them, which is of utmost importance in critical settings such as oncology and haematology.

ELIGIBILITY:
Inclusion Criteria:

* Physician or nurse in oncology or hematology
* Specialized in medical oncology or hematology

Exclusion Criteria:

* Participation to individual supervision by psycho-oncologists as part of the following training courses: CAS in psycho-oncology and course "Mieux Commu iquer"
* Participated in a study involving supervision by psycho-oncologists

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Supervisee's reflexivity (qualitative classification) | Baseline (T0) and 2 months post-baseline (i.e., T1: after the 2 months of supervision for the SPV group or 2 months waiting period for the CTRL group)
  Reflexivity will be assessed with the reflexivity indicator, a 4-level framework for classifying clinicians' narratives identified in the 5-day clinical situation recordings. This indicator has been developped in a previous study (in preparation) with the following level:
  * Level 0 - Describing: clinicians report medical and basic psychosocial facts, like a referral note.
  * Level 1 - Noticing: they mention interactions and resonate with patients' emotions but without deeper links.
  * Level 2 - Recognizing: they reflect on their interaction style, noting institutional/professional influences, and ask "what if I could do this consultation again?" to improve future practice.
  * Level 3 - Making sense: they analyze what happened, what could have been done differently, and what to do next time. Here, clinicians derive general principles, extending insights beyond the single case and shifting perspective.

SECONDARY OUTCOMES:
Feeling towards patients (questionnaire) | From supervision 1 to 4 during the 2-month intervention period (only for SPV group)
  For the SPV group only, clinicians' feelings towards presented patients will be measured with the Feeling Word Checklist (FWC; 58 items), a self-report questionnaire, prior and immediately after each supervison session. Clinicians are invited to indicate if and to what extent (5 point rating scale with 0 = not at all, and 4 = very much) the feeling described through the words are experienced regarding a given patient. We will use a translated version (french version) of the FWC.
Burnout (questionnaire) | Baseline (T0), 2 months post-baseline (T1), 3 months follow-up (FU3) and 6 months follow-up (FU6)
  The Maslach Burnout Inventory (MBI) will measure the burnout level using its 22 items divided into three scales: emotional exhaustion, depersonalization, and personal accomplishment, rated on a 6-point scale (with 0 = never, and 6 = every day). Scores for each scale are obtained by summing the responses of the corresponding items.
Supervision assessment (questionnaire) | From supervision 1 to 4 during the 2-month intervention period (only for SPV group)
  For the SPV group only, specific aspects and the overall quality of each supervision session will be assessed using a 4-item ad-hoc questionnaire completed by both the supervisee and the supervisor. The first part evaluates specific aspects of the supervision (3 items) on a 5-point Likert scale ranging from "not true at all" to "absolutely true", while the second part assesses the overall quality of the session on a 5-point scale from "unsatisfactory" to "exceptionally satisfactory". A global score, calculated by summing all responses, reflects overall satisfaction with the supervision.
  .

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatrie de liaison, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available